CLINICAL TRIAL: NCT07378943
Title: Dosing Patterns and Costs in Patients With Spinal Muscular Atrophy (SMA) Receiving Disease Modifying Therapies (DMT) - Real-world Analysis Using the Komodo Claims Data
Brief Title: A Study of Dosing Patterns and Costs in Patients With Spinal Muscular Atrophy Receiving Disease Modifying Therapies
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COAV101A1US10
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Muscular Atrophy, Spinal
Keywords: Spinal muscular atrophy; Disease modifying therapies; Real-world evidence; Dosing patterns; Treatment costs; Healthcare costs
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Nusinersen Cohort: Patients with SMA aged two years or older who received nusinersen.
- Risdiplam Cohort: Patients with SMA aged two years or older who received risdiplam.
- Onasemnogene Abeparvovec Intravenous Infusion (OAV) Monotherapy Cohort: Patients with SMA who were under two years of age and received OAV monotherapy.

SUMMARY:
The aim of this study was to assess real-world dosing patterns, long-term healthcare costs, and characteristics of SMA patients who received treatment with DMTs. DMTs included onasemnogene abeparvovec, nusinersen, and risdiplam. This study was conducted using both open and closed claims data from the Komodo Health Research Database (KRD+) between 01 January 2016 and 31 October 2024.

ELIGIBILITY:
Nusinersen and Risdiplam Cohorts:

Inclusion criteria

* Patients with ≥1 SMA diagnosis (International Classification of Diseases, Tenth Revision, Clinical Modification [ICD-10-CM] codes: G12.0, G12.1, G12.9) at any time
* Patients with ≥1 record of nusinersen or risdiplam in the data based on relevant Healthcare Common Procedure Coding System (HCPCS) codes and National Drug Code (NDC) on or after December 23, 2016
* Patients aged ≥ 2 at the index date
* Patients with ≥ 1 quarter of clinical activities within 1 year prior to the index quarter (i.e., the quarter containing the index date)
* Patients with ≥ 2 quarters of clinical activities in the first year of the follow-up

Exclusion criteria • None

Onasemnogene Abeparvovec Intravenous Infusion (OAV) Monotherapy Cohort:

Inclusion criteria

* Patients with ≥1 SMA diagnosis (ICD-10-CM codes: G12.0, G12.1, G12.9) at any time
* Patients with ≥1 record of OAV in the data based on relevant HCPCS codes and NDC on or after May 26, 2019
* Patients under 2 years old at the index date
* Patients with ≥ 2 quarters of clinical activities in their first year of follow-up

Exclusion criteria

• Treatment with nusinersen or risdiplam at any time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SMA patients with data in the KRD+ between 01 January 2016 and 31 October 2024 who received OAV, nusinersen, or risdiplam.
Sampling Method: Non-Probability Sample
Enrollment: 4114 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Patients by DMT During Each Year of DMT Treatment | Years 1, 2, 3, 4, and 5
Number of Patients Using Nusinersin During the Entire Treatment Follow-up Period | Up to 5 years
Annualized Drug and Drug Administration Costs During Each Year of Nusinersen Treatment | Years 1, 2, 3, 4, and 5
Annualized Drug and Drug Administration Costs for Nusinersen During the Entire Treatment Follow-up Period | Up to 5 years
Number of Nusinersen Injections During Each Year of Treatment | Years 1, 2, 3, 4, and 5
Number of Nusinersen Injections During the Entire Treatment Follow-up Period | Up to 5 years
Number of Patients Using Risdiplam During the Entire Treatment Follow-up Period | Up to 4 years
Annualized Drug Costs During Each Year of Risdiplam Treatment | Years 1, 2, 3, and 4
Annualized Drug Costs for Risdiplam During the Entire Treatment Follow-up Period | Up to 4 years
Annualized Risdiplam Costs Among Patients With More Than 90 Days of Supply in Year 1 | Year 1
Mean Prescribed Risdiplam Dosage During Each Year of Treatment | Year 1, 2, 3, and 4
Mean Number of Days of Supply of Risdiplam During Each Year of Treatment | Year 1, 2, 3, and 4
Mean Daily Dosage of Risdiplam During Each Year of Treatment | Year 1, 2, 3, and 4
Mean Prescribed Risdiplam Dosage During the Entire Treatment Follow-up Period | Up to 4 years
Mean Number of Days of Supply of Risdiplam During the Entire Treatment Follow-up Period | Up to 4 years
Mean Daily Dosage of Risdiplam During the Entire Treatment Follow-up Period | Up to 4 years

SECONDARY OUTCOMES:
Annualized All-cause Healthcare Costs During Each Year of OAV Follow-up | Years 1, 2, 3, and 4
  All-cause healthcare costs included costs for outpatient visits, emergency room visits, inpatient admissions, other medical visits, and pharmacy costs.
Annualized All-cause Healthcare Costs During the Entire OAV Follow-up Period | Up to 4 years
  All-cause healthcare costs included costs for outpatient visits, emergency room visits, inpatient admissions, other medical visits, and pharmacy costs.
Annualized SMA-related Healthcare Costs During Each Year of OAV Follow-up | Years 1, 2, 3, and 4
  SMA-related healthcare costs included SMA-related complications, procedures, and durable medical equipment (DME).
Annualized SMA-related Healthcare Costs During the Entire OAV Follow-up Period | Up to 4 years
  SMA-related healthcare costs included SMA-related complications, procedures, and durable medical equipment (DME).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No